CLINICAL TRIAL: NCT03683563
Title: A Prospective, Interventional Study to Investigate the Impact of Different Citrate Concentrations as Locking Solutions on Development of Biofilm and Function of Hemodialysis Catheters
Brief Title: The Impact of Different Citrate Concentrations as Locking Solutions on Development of Biofilm and Function of Hemodialysis Catheters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Bojan Medved, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CITRACOMP
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: End-Stage Kidney Disease; Renal Dialysis; Central Venous Catheter; Biofilms
Keywords: Dialysis catheters; Citrate; Locking solution
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Sodium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4% citrate (Active Comparator): dialysis catheter locked with 4% sodium citrate
  Interventions: Other: 4% sodium citrate
- 30% citrate (Experimental): dialysis catheter locked with 30% sodium citrate
  Interventions: Other: 30% sodium citrate

INTERVENTIONS:
Other: 4% sodium citrate — the catheter will be locked with 4% citrate solution after each dialysis session
  Arms: 4% citrate
Other: 30% sodium citrate — the catheter will be locked with 30% citrate solution after each dialysis session
  Arms: 30% citrate

SUMMARY:
Evidence that supports using certain concentration of trisodium citrate as a locking solution for hemodialysis catheters has not yet been established. Higher concentrations of trisodium citrate are more effective in preventing thrombosis, formation of blood clots, preventing infections and biofilm formation, but due to potential side effects, their use is limited. The aim of the study is to compare the impact of two different concentrations of tri-sodium citrate solution (30% and 4%) on the formation of biofilms in hemodialysis single-volume jugular hemodialysis catheters and to determine the effectiveness of prevention of dysfunction of hemodialysis catheters.

DETAILED DESCRIPTION:
AIM OF THE STUDY:

The aim of the study is to compare the impact of two different concentrations of trisodium citrate solution (30% and 4%) on the formation of biofilms in hemodialysis single-volume jugular hemodialysis catheters and to determine the effectiveness of prevention of dysfunction of hemodialysis catheters.

Investigators will compare the influence of two different concentrations of trisodium citrate solutions as a locking solutions for hemodialysis catheters on the formation of intraluminal biofilm, the growth of microorganisms in the lumen of the hemodialysis catheter, and the occurrence of dysfunction of hemodialysis catheters in the same patient at the same time, under the same conditions as the same length and volume of hemodialysis catheters, catheter insertion time, duration of dialysis procedures, sex, age, co-morbidity, therapy and the presence of an infection.

BACKGROUND:

The population of patients this study will include are the ones who are being treated or are supposed to start the hemodialysis treatment at the Center for Acute and Complicated Dialysis, Department for Nephrology, UKC Ljubljana and for vascular approach have newly inserted or for any reason newly replaced two single-hemodialysis catheter to the left or right inner jugular vein.

STUDY DESIGN:

The patients this study will include are the patients on chronic replacement therapy with hemodialysis, patients with acute renal failure who are on transient replacement therapy with hemodialysis and patients with renal failure starting with substitution treatment with chronic hemodialysis.

After determining the eligibility for inclusion in our study, the investigators will acquire the written consent from the patient. Patients that will be included in the study will have simultaneously inserted two jugular catheters. In the inter-dialysis period, catheters will always be filled with one catheter with 30% trisodium citrate solution, another catheter with 4% tri-sodium citrate solution.

The study will be conducted as a prospective interventional clinical trial. After dialysis, the patients' catheters will always be filled by the same protocol (one catheter with 30% trisodium citrate solution, the second catheter with 4% trisodium citrate solution). Patients will be allocated alternately between protocols 1 and 2. There are 2 protocols for filling dialysis catheters: Protocol 1: the upper (artery) catheter will be filled with 4% and lower (vein) with 30% trisodium citrate solution, Protocol 2: upper (artery) catheter will be filled with 30% and the lower (vein) with a 4% trisodium citrate solution.

Among the patients included, investigators will compare the pressure in the extracorporeal system and blood flow through dialysis catheter, time to dysfunction of hemodialysis catheters, eventual infections associated with catheter: bacteremia or sepsis, infection of the exit of dialysis catheters using different concentrations of trisodium citrate as a locking solution in the inter-dialysis period. Among the patients included, investigators will also monitor the duration of dialysis treatment, the duration of the dialysis procedure in one week, the presence of infection, age, co-morbidity, concomitant therapy (treatment with anticoagulation and anti-aggregation drugs, the presence of immunosuppression, antibiotics). In approximately 5 patients we will simultaneously remove the dialysis catheter due to any medical indication and then via an electronic microscope and stereomicroscope evaluate morphological characteristics of biofilm. Investigators will also evaluate the microbiological characteristics of biofilms using microbiological methods.

EXPECTED RESULTS:

It is expected that the occurrence of dysfunction or the number of catheter days in the same patients using different concentrations of trisodium citrate solutions in inter-dialysis period will be statistically different.

It is expected that the morphological parameters of biofilm will be statistically different using different concentration solution of trisodium citrate (30%, 4%). It is also expected that the microbiological characteristics of biofilm will differ according to the used concentration of the trisodium citrate solution in the inter-dialysis period.

The data investigators will receive can help to understand the adverse events occurring with the use of hemodialysis catheters, filling with different concentrations of trisodium citrate solutions.

ELIGIBILITY:
Inclusion Criteria:

* CKD on dialisys
* AKI on dialisys

Exclusion Criteria:

* systemic bacterial infection at the time of catheter insertion
* local infection at the catheter insertion site
* hypersensitivity to citrate
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
catheter dysfunction | within 6 months after catheter insertion
  occurrence of dysfunction of dialysis catheter (expressed as catheter days)

SECONDARY OUTCOMES:
identification of microorganisms | an average of 1 year
  investigators will identify potential microorganisms on the surfaces of the hemodialysis catheter by method "sonication" of the catheter segment and afterward cultivation in solid and liquid media
distribution of biofilm | an average of 1 year
  investigators will inspect distribution of biofilm (% area) along inner surface of the dialysis catheter by electronic microscope

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided